CLINICAL TRIAL: NCT00714142
Title: Renal Blood Flow Measurement With PET
Brief Title: Renal Blood Flow Measurement With Positron Emission Tomography (PET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jeffrey L. Lacy (Industry)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor-Investigator, Jeffrey L. Lacy, President, Proportional Technologies, Inc.
Organization: Proportional Technologies, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UW HS IRB 2008-0097; DK58466
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Renal Failure; Renal Artery Stenosis
Keywords: Renal blood flow; PET imaging
MeSH Terms: conditions — Renal Insufficiency; Renal Artery Obstruction | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Normal volunteers
  Interventions: Drug: 62Cu-ethylglyoxal bis(thiosemicarbazone); Drug: 15O-water; Procedure: Positron Emission Tomography
- 2 (Active Comparator): Renal failure patients on dialysis
  Interventions: Drug: 62Cu-ethylglyoxal bis(thiosemicarbazone); Drug: 15O-water; Procedure: Positron Emission Tomography
- 3 (Active Comparator): Renal artery stenosis patients
  Interventions: Drug: 62Cu-ethylglyoxal bis(thiosemicarbazone); Drug: 15O-water; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: 62Cu-ethylglyoxal bis(thiosemicarbazone) — 15-25 mCi, IV
Drug: 15O-water — 10-20 mCi, IV
Procedure: Positron Emission Tomography — PET Scan

SUMMARY:
Two investigational chemical tracers, 62Cu-ethylglyoxal bis(thiosemicarbazone) (62Cu-ETS) and 15O-water, will be used in this study to look at how blood moves through the kidneys. The purpose of the study is to see if 62Cu-ETS is effective in showing the blood supply to the kidneys compared to 15O-water. The tracer mixes with the blood and moves through the body. Using positron emission tomography (PET scan) the researchers can see the tracer and can learn more about how the blood moves through the kidneys. The study invites participants who are healthy, without any heart or kidney disease, patients who have kidney disease that require dialysis, and patients who may have a blockage in one of the arteries supplying blood to the kidneys.

ELIGIBILITY:
Arm 1.

Inclusion Criteria:

* males and females, age 18-40 years
* willingness to provide written informed consent

Exclusion Criteria:

* history of coronary artery disease (CAD)
* history of renal disease
* risk factors for cardiac disease, renal disease, or atherosclerosis, including diabetes mellitus, hypertension, tobacco abuse, hyperlipidemia, family history of CAD or chronic renal failure
* history of liver disease or other significant disease
* pregnant females

Arm 2.

Inclusion Criteria:

* males and females, age > 18 years
* active hemodialysis or peritoneal dialysis for at least six months
* any etiology of chronic renal failure except active glomerular nephritis
* presence of two kidneys
* willingness to provide written informed consent

Exclusion Criteria:

* decompensated heart failure (subjects must be on stable medical therapy for one month)
* any previous renal transplant (subjects may be on renal transplant waiting list)
* history of liver disease
* pregnant females

Arm 3.

Inclusion Criteria:

* males and females, age > 18 years
* documented evidence of renal artery stenosis equivalent to a 75% stenosis by one of the following clinical tests: MRA, Doppler, Renal Angiogram, Abnormal captopril renal scan
* evidence of renal insufficiency with serum creatinine >= 1.3 mg/dL
* presence of two kidneys
* willingness to provide written informed consent

Exclusion Criteria:

* revascularization of stenotic renal artery
* decompensated heart failure (subjects must be on stable medical therapy for one month)
* any previous renal transplant (subjects may be on renal transplant waiting list)
* history of liver disease
* pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Obtain preliminary information on efficacy for quantification of regional renal perfusion in two target clinical populations with a full range of renal disease using 150-water PET and 62Cu-ETS PET | one day

SECONDARY OUTCOMES:
Assess the safety of the drug 62Cu-ETS through expansion to two target patient populations and increase the size of the normal subjects group | one day

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Lacy, PhD, Principal Investigator — Proportional Technologies, Inc.; Charles K Stone, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States